CLINICAL TRIAL: NCT06236373
Title: The Unmet Needs of Cancer Survivors in Ausl IRCCS Reggio Emilia Reality: a Qualitative Study and Framework Analysis
Brief Title: The Unmet Needs of Cancer Survivors in Ausl IRCCS Reggio Emilia
Acronym: Survivorship
Status: Recruiting | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Azienda USL - IRCCS di Reggio Emilia (Unknown)
Responsible Party: Principal Investigator, Stefania Costi, PhD, University of Modena and Reggio Emilia
Other Study IDs: UN2023
Record Dates: First submitted 2024-01-10; First posted 2024-02-01 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Breast Cancer; Prostate Cancer; Thyroid Cancer; Colorectal Cancer; Lymphoma; Multiple Myeloma; Neoplasms
Keywords: Unmet needs; Quality of Life; Survivorship care; Cancer; Survivors; Care givers; Stakeholder; Breast; Prostate; Thyroid; Colorectal; Myeloma
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Thyroid Neoplasms; Colorectal Neoplasms; Lymphoma; Multiple Myeloma; Thyroid Diseases; Neoplasms, Plasma Cell | interventions — Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cancer Survivors: Cancer Survivors
  Interventions: Other: Focus Groups or Interviews
- Cancer Survivors Caregiver: Family members or/and caregivers
  Interventions: Other: Focus Groups or Interviews
- Cancer Survivors Stakeholders: Health professionals, patients associations
  Interventions: Other: Focus Groups or Interviews

INTERVENTIONS:
Other: Focus Groups or Interviews — Focus groups and qualitative interview will be conducted with patients, caregivers and stake-holders trying to identify unmet needs of cancer survivors after the acute treatment phase. Individual interviews (in presence or online) will be hold as alternative if it will not be possible (due to logistical or personal problems) to participate in a focus group or if the number of people who would have agreed to participate in that focus group is less than 3

SUMMARY:
This qualitative study seeks to explore the unmet needs of individuals who have recently undergone a cancer diagnosis and completed the acute phase of treatment. The primary objective is to utilize the experiences of patients, caregivers, and stakeholders to enhance the aftercare provided to cancer survivors. By delving into patient perceptions regarding unmet needs in cancer aftercare, the study aims to identify areas for redesigning and improving services to minimize these needs and ultimately enhance patient outcomes. Importantly, the investigation incorporates insights from patients, their caregivers, and stakeholders.

The research will employ qualitative methods, specifically focus groups and interviews, to gather comprehensive perspectives from individuals in the Ausl IRCCS Reggio Emilia district who have completed treatment for breast, prostate, colorectal, thyroid, and multiple myeloma cancers. Including patients with diverse cancer types is crucial for capturing a broad spectrum of experiences.

During data collection, both focus group discussions and interviews will be recorded in audio format and transcribed verbatim. This meticulous approach ensures an accurate representation of participants' voices and experiences. The subsequent analysis will employ a combination of framework and thematic analysis to extract meaningful insights and synthesize the data effectively.

The study's ultimate goal is to leverage the findings to optimize aftercare services for cancer survivors within the local context of Ausl IRCCS Reggio Emilia. By incorporating the perspectives of patients, caregivers, and stakeholders, the research aims to contribute valuable insights that can inform the redesign and improvement of aftercare services, ultimately benefitting cancer survivors in the region.

DETAILED DESCRIPTION:
The escalating global population of cancer survivors (CSs) underscores the imperative to offer services tailored to address their specific unmet needs. Individuals are designated as 'cancer survivors' from the moment of diagnosis onward throughout their lifetime. Despite this, there is a worldwide acknowledgment that CSs encounter a spectrum of physical, psychosocial, spiritual, informational, and practical challenges, often leading to unmet needs that frequently go unrecognized and unaddressed.

Unmet needs, in this context, refer to those requirements perceived by individuals as lacking the necessary level of service for achieving optimal well-being. These can be characterized as unsatisfied needs for which CSs desire additional assistance or support. A profound comprehension and measurement of CSs' unmet needs play a pivotal role in identifying gaps in their care experiences, providing an opportunity to deliver patient-centered services.

Effective care delivery not only enhances patient outcomes and quality of life but also contributes to increased satisfaction with care. This, in turn, may lead to a reduced demand for health and social care services. The qualitative study outlined here seeks to delve into the unmet needs of individuals who have undergone a cancer diagnosis within the past years and have completed the acute phase of treatment.

The study aims to leverage the experiences of patients, caregivers, and stakeholders to optimize cancer survivorship care. Specifically, the investigation will focus on the unmet needs of cancer survivors post the acute treatment phase for some of the most prevalent forms of cancer with a life expectancy of at least five years.

Namely:

1. To investigate the unmet needs perceived by cancer survivors in AUSL IRCCS Reggio Emilia setting.
2. To determine the area of impact on health encompassed by those unmet needs to create a direct link to the ICF.
3. To determine which Patient Reported Outcome Measure aimed at identifying cancer survivors' unmet needs will best investigate those ICF components connected to common cancer survivors' unmet needs to implement it in their routine assessment.
4. To identify the services that need to be implemented to provide support to the true needs of local cancer survivors.
5. To develop a Survivorship care plan model coherent with patients' expectations and health care system economic resources.

Utilizing focus groups and interviews, the research will recruit participants from the AUSL - IRCCS Reggio Emilia district who have completed treatment for breast, prostate, colorectal, thyroid, and multiple myeloma cancers. The study will adhere to a structured schedule for conducting focus groups and interviews, accommodating participants in individual interviews if logistical or personal challenges arise.

Each focus group, homogeneous in terms of pathology, will include 4 to 8 participants, with a total ranging between 30 and 60 participants based on Krueger's recommendations. Audio recording and verbatim transcription of focus groups and interviews will facilitate subsequent framework and thematic analysis to extract meaningful insights.

The study's objectives encompass investigating perceived unmet needs, determining the health impact linked to these needs within the International Classification of Functioning, Disability, and Health (ICF), identifying suitable Patient Reported Outcome Measures, pinpointing services for implementation, and developing a Survivorship care plan model aligning with patient expectations and healthcare system resources.

The focus groups and interviews, including patients with or without linked caregivers, will be systematically transcribed and analyzed using framework and thematic analysis methodologies.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged18 years or over.
* Individuals who have a history of breast, prostate, thyroid, colorectal, multiple myeloma or lymphoma cancer within the past years who have completed the acute phase of treatment, and are in follow-up or are receiving maintenance treatment;
* Caregivers for an individual who meets the above criteria, who are aged 18 years or over.
* Stakeholders for individual who meets the above criteria, who are aged 18 years or over.

Exclusion Criteria:

* Individuals who do not wish to participate
* Individuals who do not understand and/or speak Italian
* Individuals with significant cognitive impairment, learning difficulty, or communication difficulty such that understanding the nature of the study, the interview questions, or participating in a focus group or an on-line or in-presence interview would not be practical.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer survivors who have recived a diagnosis of the following types of cancer:
  * breast,
  * prostate,
  * thyroid,
  * colorectal,
  * multiple myeloma
  * lymphoma
  Or caregiver/stakeholder of an individual who meets the inclusion criteria and are aged 18 years or over
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Experience of Self-reported perception of Unmet Needs | 1- In the last three months 2- In the last 12 months
  Evaluation from the patients' point of view on their perception of unmet needs, which are those needs that lack the level of service an individual perceives as necessary to achieve optimal well-being. Semi-structured qualitative interviews will be conducted with patients' participating in the study to collect information and description of unsatisfied needs for which cancer survivors would like to receive more assistance or support. These may include (as an example): Stress or other psychological demands, Informational needs, Physical needs, Spiritual needs, among others.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Costi, PhD, Principal Investigator — Physical Medicine and Rehabilitation Unit, Azienda Unità Sanitaria Locale - IRCCS di Reggio Emilia
Locations (1):
- Casa della Salute ex Spallanzani, Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Recording will be anonymised and transcripted verbatim. This anonimised material could be shared with other researchers on request

REFERENCES:
- [Background] Contri A, Paltrinieri S, Torreggiani M, Chiara Bassi M, Mazzini E, Guberti M, Campanini I, Ghirotto L, Fugazzaro S, Costi S. Patient-reported outcome measure to implement routine assessment of cancer survivors' unmet needs: An overview of reviews and COSMIN analysis. Cancer Treat Rev. 2023 Nov;120:102622. doi: 10.1016/j.ctrv.2023.102622. Epub 2023 Sep 9. PMID 37713972
- [Background] Tralongo P, McCabe MS, Surbone A. Challenge For Cancer Survivorship: Improving Care Through Categorization by Risk. J Clin Oncol. 2017 Oct 20;35(30):3516-3517. doi: 10.1200/JCO.2017.74.3450. Epub 2017 Aug 23. No abstract available. PMID 28834437
- [Background] Santos ATCD, Silva RPD, Almeida LM, Bosi MLM, Menezes MFB, Skaba MMVF, Nigenda G, Arruda CAM, Pinheiro CPO, Gonzalez-Robledo MC, Knaul FM. Cancer survivorship needs in Brazil: Patient and family perspective. PLoS One. 2020 Oct 8;15(10):e0239811. doi: 10.1371/journal.pone.0239811. eCollection 2020. PMID 33031426
- [Background] Nekhlyudov L, Mollica MA, Jacobsen PB, Mayer DK, Shulman LN, Geiger AM. Developing a Quality of Cancer Survivorship Care Framework: Implications for Clinical Care, Research, and Policy. J Natl Cancer Inst. 2019 Nov 1;111(11):1120-1130. doi: 10.1093/jnci/djz089. PMID 31095326
- [Background] McCanney J, Winckworth-Prejsnar K, Schatz AA, Nardi EA, Dwyer AJ, Lieu C, Biru Y, Carlson RW. Addressing Survivorship in Cancer Care. J Natl Compr Canc Netw. 2018 Jul;16(7):801-806. doi: 10.6004/jnccn.2018.7054. PMID 30006422
- [Derived] Contri A, Ghirotto L, Cavuto S, Schiavi M, Cervi E, Soffientini V, Soncini S, Botti S, Frasoldati A, Torreggiani M, Costi S. From patient voices to optimal PROMs: a mixed methods framework for cancer survivorship care. J Cancer Surviv. 2025 Nov 7. doi: 10.1007/s11764-025-01899-x. Online ahead of print. PMID 41201742
- [Derived] Contri A, Costi S, Guberti M, Soncini S, Botti S, Frasoldati A, Torreggiani M, Ghirotto L. Voices of Survivorship: The Unmet Needs of Italian Cancer Survivors. A Qualitative Study. Cancer Med. 2025 Aug;14(15):e71121. doi: 10.1002/cam4.71121. PMID 40747540